CLINICAL TRIAL: NCT02719769
Title: Evaluation of Clinical Performance of the Accelerate ID/AST System for Positive Blood Culture Identification & Antimicrobial Susceptibility Testing
Brief Title: Clinical Performance of the Accelerate ID/AST System for Positive Blood Culture
Status: Completed | Type: Observational
Sponsor: Accelerate Diagnostics, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CP000004; CP00002 (Other: Accelerate Diagnostics)
Record Dates: First submitted 2016-01-11; First posted 2016-03-25 (Estimated); Last update posted 2017-09-27 (Actual); Status verified 2017-09

CONDITIONS: Bacteremia; Fungemia
Keywords: Positive Blood Culture
MeSH Terms: conditions — Bacteremia; Fungemia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Frozen positive blood cultures and bacterial and yeast isolates
Oversight: Data Monitoring Committee: No

SUMMARY:
The "Evaluation of Clinical Performance of the Accelerate ID/AST System for Positive Blood Culture Identification & Antimicrobial Susceptibility Testing" is designed to validate the clinical performance of the Accelerate ID/AST System for positive blood culture identification and susceptibility testing in a clinical setting. The data from this study will be used to support the 510(k) submission for FDA clearance and global registrations of the device intended for in vitro diagnostic use.

DETAILED DESCRIPTION:
The clinical study entitled "Evaluation of Clinical Performance of the Accelerate ID/AST System for Positive Blood Culture Identification & Antimicrobial Susceptibility Testing" is designed to demonstrate the clinical performance of the Accelerate ID/AST System for positive blood culture identification (ID) and antimicrobial susceptibility testing (AST) in a clinical setting compared to reference results. Approximately 3,000 positive blood culture samples (across all Clinical Sites) will be tested on the investigational device and reference methods. Up to 50% of samples enrolled will be comprised of seeded blood cultures prepared from clinical stock isolates. Quality Control testing will be performed each day of testing. The study population is comprised of left-over clinical specimens that are indicated as positive by blood culture monitoring systems utilized by clinical microbiology laboratories. Positive blood culture samples must be tested on the Accelerate ID/AST System within 8 hours of positivity by the blood culture monitoring system. Testing of clinical samples will continue until the required sample size for each target organism and antimicrobial agent, including sufficient on-scale and resistant strains, are tested across all the sites.

ELIGIBILITY:
Inclusion Criteria:

* De-identified positive blood culture specimens (6 mL aliquot)
* Seeded blood culture specimens (stock) from archived bacterial and yeast isolates

Exclusion Criteria:

* Sample volume available < 6 mL
* Positive Blood Culture sample > 8 hours post-positivity
* Sample from patient previously enrolled
* Sample from blood culture media that contain charcoal e.g., BACTAlert FA, FN bottles
* Samples from Mycobacterial-type blood culture media e.g., BACTEC Myco/F Lytic, BacT/ALERT MP Bottle, VersaTREK Myco

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Clinical specimens that are indicated as positive by blood culture monitoring systems utilized by clinical microbiology laboratories.
Sampling Method: Non-Probability Sample
Enrollment: 4009 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2016-05 (Actual); Study Completion 2017-01-12 (Actual)

PRIMARY OUTCOMES:
Comparison Study - ID Performance | Approximately 9 months (including pre-clinical phase)
  Positive and Negative Percent Agreement with Comparator Method (Vitek2) by Bacterial/Fungal Target

SECONDARY OUTCOMES:
Comparison Study - AST Performance | Approximately 9 months (including pre-clinical phase)
  Essential and Categorical Agreement with CLSI Frozen Reference Method (BMD) by Antimicrobial

CONTACTS AND LOCATIONS:
Overall Officials: Constance Bridges, B.S., MBA, Principal Investigator — Accelerate Diagnostics, Inc.
Locations (14):
- United States (14):
  - Banner Health- Laboratory Sciences of Arizona, Gilbert, Arizona
  - Accelerate Diagnostics Inc., Tucson, Arizona
  - UCLA Medical Center, Los Angeles, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - MRI Global, Palm Bay, Florida
  - Loyola University Medical Center, Maywood, Illinois
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Johns Hopkins University School of Medicine, Baltimore, Maryland
  - Mayo Clinic, Rochester, Minnesota
  - Lab Alliance of Central New York LLC, Liverpool, New York
  - The Ohio State University, Columbus, Ohio
  - Geisinger Clinic, Danville, Pennsylvania
  - med fusion LLC, Lewisville, Texas
  - Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No